CLINICAL TRIAL: NCT00054756
Title: Study of Thyrotropin Releasing Hormone in Patients With Thyroid or Pituitary Abnormalities
Brief Title: Study of Thyrotropin-Releasing Hormone in Normal Volunteers and in Patients With Thyroid or Pituitary Abnormalities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 030098; 03-DK-0098 (Other: NIHCC)
Record Dates: First submitted 2003-02-07; First posted 2003-02-10 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-04

CONDITIONS: Healthy; Pituitary Disease; Thyroid Disease
Keywords: Hypothalamic Releasing Factor; Neuropeptide; Diagnostic Testing; Pituitary Tumors; Central Hypothyroidism; Pituitary Disorder; Thyroid Disorder; Healthy Volunteer
MeSH Terms: conditions — Pituitary Diseases; Thyroid Diseases; Pituitary Neoplasms; Hypothyroidism | interventions — Thyrotropin-Releasing Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Thyrotropin Releasing Hormone (Experimental): Subjects receiving TRH (Thyrotropin Releasing Hormone)
  Interventions: Drug: TRH (Thyrotropin Releasing Hormone)

INTERVENTIONS:
Drug: TRH (Thyrotropin Releasing Hormone)

SUMMARY:
This study will determine the safety and activity of a new formulation of thyrotropin-releasing hormone (TRH), a drug used for diagnosing and evaluating patients with certain thyroid gland abnormalities. Normal thyroid gland function depends on proper chemical signaling between the thyroid gland, the hypothalamus (the part of the brain where TRH is made), and the pituitary (another part of the brain). The TRH test helps assess this interaction. Production of the only FDA-approved preparation of TRH was stopped in July 2002. As a result, to have a continuous source of TRH available for NIH clinical and research purposes, the NIH Clinical Center (CC) Pharmacy Department produced a pharmaceutical grade formulation of TRH for patient use. This study will test the CC formulation in healthy volunteers to show that its activity and side effects are similar to those of the previously available commercial test preparation. It will then be studied in CC patients for whom the diagnostic test is recommended.

Healthy volunteers between 18 and 65 years of age and all patients requiring TRH evaluation of hypothalamic-pituitary-thyroid gland interaction may be eligible for this study. Patients include those with pituitary reserve, inconsistent thyroid function test, inappropriate TSH secretion, or pre- and post-operative evaluation of pituitary tumors. Normal volunteers will be screened with a medical history, physical examination, and blood tests. Women of child-bearing potential will be given a pregnancy test; pregnant and breast-feeding women may not participate.

The TRH test procedure will be the same for healthy volunteers and patients. All participants fast from midnight before the morning of the test. In the morning, a catheter (flexible plastic tube) is inserted into an arm vein for easy injection of the TRH and collection of blood samples. Blood pressure is monitored before and during the test. A blood sample is drawn, and then TRH is given through the catheter over a 1-minute period. Another nine blood samples are collected over a 3-hour period from the time of the TRH injection for measuring levels of various hormones. A total of less than 4 tablespoons of blood is taken for the test.

DETAILED DESCRIPTION:
Thyrotropin releasing hormone (TRH) is a neuropeptide used in the diagnostic evaluation of patients with dysfunction of the hypothalamic-pituitary-thyroid (HPT) axis. In healthy individuals, administration of TRH intravenously results in pituitary secretion of thyrotropin [thyroid-stimulating hormone (TSH)], which in turn stimulates the thyroid gland release of thyroid hormones; thyroxine (T4) and triiodothyronine (T3). TRH stimulates the secretion of other pituitary hormones under normal physiologic as well as pathologic conditions.

Under this protocol, TRH is used for routine diagnostic testing and research studies in adults and children. It is produced by the Pharmaceutical Development Section of the Clinical Center Pharmacy at the NIH. The safety, activity and comparability of this preparation were demonstrated in a small group of normal volunteers prior to its release for diagnostic and research use.

ELIGIBILITY:
* DIAGNOSTIC STUDY PROTOCOL

Inclusion Criteria:

-All adults and children requiring dynamic testing of the hypothalamic-pituitary axis for the evaluation of pituitary reserve, inconsistent thyroid function test, inappropriate TSH secretion, or pre-and post-operative evaluation of pituitary adenomas (glycoprotein hormone secreting tumors, growth hormone secreting tumors and TSH secreting tumors).

Exclusion Criteria:

* Uncontrolled hypertension;
* Uncontrolled seizure disorder;
* Unstable coronary disease;
* Known allergy to TRH.

RESEARCH PROTOCOLS

-TRH is available for use in other IRB approved research protocols either using the standard diagnostic testing protocol or the modified TRH test.

Exclusion Criteria:

* Untreated hypertension;
* Coronary artery disease;
* History of asthma;
* History of seizures;
* Pregnancy;
* Known allergy to TRH.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2003-02-07; Primary Completion 2014-09-26 (Actual); Study Completion 2014-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Klubo-Gwiezdzinska, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jackson IM. Thyrotropin-releasing hormone. N Engl J Med. 1982 Jan 21;306(3):145-55. doi: 10.1056/NEJM198201213060305. No abstract available. PMID 6798440
- [Background] Haigler ED Jr, Pittman JA Jr, Hershman JM, Baugh CM. Direct evaluation of pituitary thyrotopin reserve utilizing synthetic thyrotopin releasing hormone. J Clin Endocrinol Metab. 1971 Oct;33(4):573-81. doi: 10.1210/jcem-33-4-573. No abstract available. PMID 4999252
- [Background] Faglia G. The clinical impact of the thyrotropin-releasing hormone test. Thyroid. 1998 Oct;8(10):903-8. doi: 10.1089/thy.1998.8.903. PMID 9827657
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-DK-0098.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thyrotropin Releasing Hormone
Started | 96
Completed | 94
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Thyrotropin Releasing Hormone
Number analyzed (Participants) | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 92
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 38 [9 to 75]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants did not report sex.
  Participants
    number analyzed (Participants) | 94
    Female | 58
    Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 19
  White | 68
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: TSH Response to TRH
Description: Serum TSH Levels in Response to TRH Administration
Time Frame: 180 minutes from infusion
Population: 2 participants did not have results drawn at 180 minutes
Measure: Mean (Full Range); unit: mcIU/mL
Arm/Group | Thyrotropin Releasing Hormone
Number analyzed (Participants) | 94
mcIU/mL | 11.47 [0.01 to 233]

ADVERSE EVENTS:
Time Frame: 180 minutes after injection of TRH
Arm/Group | Thyrotropin Releasing Hormone
All-Cause Mortality (participants affected / at risk) | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96
Other Adverse Events (participants affected / at risk) | 0/96

LIMITATIONS AND CAVEATS:
This study was conducted under an IND because the TRH was produced at NIH after the FDA approved manufacturer stopped producing the product. The intent of the study was to provide TRH for diagnostic purposes for patients at the NIH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes